CLINICAL TRIAL: NCT02801318
Title: Role of REM Sleep Alterations in Post Operative Delirium After Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DELI-SLEEP
Record Dates: First submitted 2015-07-16; First posted 2016-06-15 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Delirium Symptoms
Keywords: Patient

ARMS (1):
- Polysomnography (Other)
  Interventions: Procedure: Polysomnography

INTERVENTIONS:
Procedure: Polysomnography

SUMMARY:
Acute confusional states known as delirium frequently occur in Intensive Care Units (ICU), mostly after cardiac surgery, leading to serious consequences. Sleep deprivation has been described in ICU patients and is considered as a risk factor for delirium but its role is still unknown. It is therefore essential to identify whether sleep deprivation and more specifically REM sleep alterations could facilitate occurence of delirium in ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had a cardiac surgery with extracorporeal circulation.
* Patients who were extubated at Day 0.
* Patients without any operation or anesthetic complication.
* Patients who speak French.
* Patients without TNC at Day 1.
* Patients who had completed the questionnaires before operation.

Exclusion Criteria:

* Age < 18 years old.
* Delirium at Day 1.
* Central nervous system pathology or psychiatric pathology known and treated.
* Concomitant use of neuropsychiatric treatment before surgery that interferes with sleep.
* Clinical condition alteration before polysomnography exam.
* Continue sedation required before Day 3 polysomnography exam.
* Agitation or clinical alteration that did not allow Day 3 polysomnography exam.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Primary Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
significant difference of REM sleep quantity in polysomnography at day 3 | Day 3